CLINICAL TRIAL: NCT02704182
Title: Role of Transcranial Direct Current Stimulation (tDCS) in Reduction of Pain and Postsurgical Opioid Consumption in Total Knee Arthroplasty (TKA)
Brief Title: Transcranial Direct Current Stimulation for Postoperative Pain in Knee Arthroplasty
Acronym: TDCSTKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS in TKA
Record Dates: First submitted 2016-01-31; First posted 2016-03-09 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Knee Replacement
Keywords: Arthroplasties, Knee Replacement
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real tDCS (Active Comparator): Direct current stimulation using anodal electrode, 25 patients received real anodal tDCS on the motor area for 20 minutes every day for 4 consecutive days.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Sham direct current stimulation, 25 patients received sham anodal tDCS on the motor area for 20 minutes every day for 4 consecutive days.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — 25 patients received real anodal tDCS on the motor area for 20 minutes every day for 4 consecutive days.
  Arms: Real tDCS
Device: Sham tDCS — 25 patients received sham anodal tDCS on the motor area for 20 minutes every day for 4 consecutive days.
  Arms: Sham tDCS

SUMMARY:
The objective of this study is to detect the effect of trans-cranial direct current stimulation on postoperative pain and opioid consumption in total knee arthro-plasty patients. Fifty patients undergoing unilateral TKA will be randomly assigned to receive 4 sessions, total of 80 minutes of real (n=25) or sham tDCS (n=25). Stimulation will be given on 4 consecutive postoperative days, group 1 will receive real stimulation with the active electrode over the leg representation of the motor strip (cortical motor area of the leg) and the reference electrode over the arm, group 2 will receive Sham tDCS. Pain level will be evaluated according to visual analogue scale (VAS) and LANSS pain scale before (base line) after 1st, 2nd, 3rd and 4th sessions.

DETAILED DESCRIPTION:
The study aims to to detect the effect of trans-cranial direct current stimulation on postoperative pain and opioid consumption in total knee arthro-plasty patients.

Fifty patients undergoing unilateral TKA will be randomly assigned to receive 4 sessions, total of 80 minutes of real (n=25) or sham tDCS (n=25). Stimulation will be given on 4 consecutive postoperative days, group 1 will receive real stimulation with the active electrode over the leg representation of the motor strip (cortical motor area of the leg) and the reference electrode over the arm, group 2 will receive Sham tDCS.

Pain level will be evaluated according to visual analogue scale (VAS) and LANSS pain scale before (baseline) after 1st, 2nd, 3rd and 4th sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Providing informed consent to participate in the study.
2. age >30 years and <60 years both genders.
3. ASA I to II patients.
4. postoperative unilateral total knee arthroplasty.

Exclusion Criteria:

1. Contraindications to transcranial brain stimulation: presence of a history of epilepsy, implantable devices (ventriculo-peritoneal shunts, pacemakers, intracranial metal implants).
2. Neurological or psychiatric pathology.
3. Patients taking major centrally acting drugs (anti-epileptics or antidepressants) or high-dose opioid.
4. History of substance abuse.
5. Severe cardio-pulmonary, renal, hepatic diseases.
6. Pregnancy and lactation.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Opioids consumption per 24 hours at the 4th day postoperative | day 4 postoperative
  Measuring the consumption dose of opioids per 24 hours at the fourth day
Opioids consumption / 24 hours at the third day postoperative | day 3 postoperative
  Measuring the consumption dose of opioids per 24 hours at the third day postoperative
Opioids Consumption / 24 hours at the second day postoperative | day 2 postoperative
  Measuring the consumption dose of opioids per 24 hours at the second day post-operative
Opioids consumption / 24 hours at the 1st day postoperative | 1st day postoperative
  Measuring the consumption dose of opioids per 24 hours at the 1st day postoperative

SECONDARY OUTCOMES:
Opioid side effects | 4th post operative day
  Record Opioid-related adverse effects (nausea and/or vomiting and the need for alizapride 50mg IV).
Pain assessment by VAS | 3rd postoperative day
  Pain Assessment using Visual Analogue Scale
Pain assessment by VAS | 2nd postoperative day
  Pain Assessment using Visual Analogue Scale
Pain assessment by VAS | 1st postoperative days
  Pain Assessment using Visual Analogue Scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khedr EM, Sharkawy ESA, Attia AMA, Ibrahim Osman NM, Sayed ZM. Role of transcranial direct current stimulation on reduction of postsurgical opioid consumption and pain in total knee arthroplasty: Double randomized clinical trial. Eur J Pain. 2017 Sep;21(8):1355-1365. doi: 10.1002/ejp.1034. Epub 2017 Apr 25. PMID 28440034